CLINICAL TRIAL: NCT03781440
Title: Regional Anesthesia for Cardiothoracic Enhanced Recovery for Patients Undergoing Cardiac Surgery Via Sternotomy
Brief Title: Regional Anesthesia for Cardiothoracic Enhanced Recovery
Acronym: RACER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Chi-Ho Ban Tsui, Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 47647
Record Dates: First submitted 2018-12-18; First posted 2018-12-19 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Opioid Use; Anesthesia, Local; Cardiac Disease; Pain, Acute
MeSH Terms: conditions — Heart Diseases; Acute Pain | interventions — Lidocaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bilateral ESP catheter with Lidocaine (Experimental): All participants will get the Erector Spinae Plane (ESP) catheters. Prior to transfer to the operating room, participants will receive bilateral ESP catheters at T7 level under ultrasound guidance. This arm is the treatment group and will receive lidocaine via alternating side automated infusion pump bolus dosing, continued until chest tube removal or postoperative day 5 (whichever occurs earliest).
  Interventions: Procedure: Bilateral ESP catheter with lidocaine
- Bilateral ESP catheter with saline (Placebo Comparator): All participants will get the Erector Spinae Plane (ESP) catheters. This arm is the control group and will have normal saline administered via ESP catheters, continued until chest tube removal or postoperative day 5 (whichever occurs earliest).
  Interventions: Procedure: Bilateral ESP catheter with saline

INTERVENTIONS:
Procedure: Bilateral ESP catheter with lidocaine — All participants will get the Erector Spinae Plane (ESP) catheters. Prior to transfer to the operating room, participants will receive bilateral ESP catheters at T7 level under ultrasound guidance. This arm is the treatment group and will receive lidocaine via alternating side automated infusion pump bolus dosing, continued until chest tube removal or postoperative day 5 (whichever occurs earliest).
  Arms: Bilateral ESP catheter with Lidocaine
Procedure: Bilateral ESP catheter with saline — All participants will get the Erector Spinae Plane (ESP) catheters. This arm is the control group and will have normal saline administered via ESP catheters, continued until chest tube removal or postoperative day 5 (whichever occurs earliest).
  Arms: Bilateral ESP catheter with saline

SUMMARY:
The erector spinae plane block (ESPB) is a novel regional analgesic technique that provides pain relief with a peripheral nerve block catheter. The goal of this study is to see if bilateral ESPB catheters can improve clinical outcomes in patients undergoing cardiac surgery via sternotomy, such as decreasing the duration of postoperative mechanical ventilation, need for intravenous opioid medications, length of stay in the intensive care unit (ICU), and improving pain scores.

ELIGIBILITY:
Inclusion Criteria:

* Give consent to participate in study
* planned sternotomy
* specific procedures: CABG (coronary artery bypass grafting) or AVR (aortic valve repair or replacement) or MVR (mitral valve repair or replacement) or combination of any of 2 of these
* Primary or first redo sternotomy

Exclusion Criteria:

* Participants who cannot give consent
* Patients who are clinically unstable or require urgent/emergent intervention
* more than1 prior sternotomy
* planned aortic arch procedures
* preoperative coagulopathy (INR >1.5, PTT >35) or ongoing anticoagulation (heparin infusion, therapeutic low molecular weight heparin, warfarin, dual antiplatelet therapy)
* Severe ventricular dysfunction (left or right ventricle)
* Symptomatic heart failure (systolic or diastolic)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Opioid Consumption | Duration of postoperative recovery (typically 1-2 weeks)
  IV and PO opioid requirements converted to morphine equivalent

SECONDARY OUTCOMES:
Delirium and agitation post-operatively | Duration of ICU stay (typically 2-5 days)
  Richmond Agitation-Sedation Score from -5 to +4 (-5 is the most sedation, +4 is the least sedated.
Determine post-operative pain scores | Duration of postoperative recovery (typically 1-2 weeks)
  11-point numerical rating scale (NRS) from 0-10, 0 signifying no pain, 10 signifying the worse pain.
Median time to extubation in patients with ESPB | Duration of postoperative recovery (typically 1-2 weeks)
  duration in mechanical ventilation in hours
Length of stay in hospital | Duration of postoperative recovery (typically 1-2 weeks)
  number of post-operative days spent in hospital
Length of stay in ICU | Duration of postoperative recovery (typically 1-2 weeks)
  number of post-operative days spent in ICU
Quality of recovery at 72 hours | post-operative day 3
  Survey based (Quality of Recover 15) patient reported outcomes. There are 15 questions based on a scale of 0-10 per questions, 0 signifying the worst outcome, 10 signifying the best, for a score range of 0-150.
Inflammatory biomarker analysis | First panel pre-incision; second panel 6hrs (+/-3hrs) post-procedure; third panel 24hrs (+/-3hrs) post-procedure; fourth panel 48hrs (+/-3hrs) post-procedure
  Pro and anti-inflammatory biomarker panel at 4 time points perioperatively. We will be analyzing IL10 concentrations as an anti-inflammatory biomarker and IL6 and TN alpha as pro-inflammatory biomarkers in either a ELISA assay or Luminex.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Brodt, MD, Principal Investigator — Stanford University; Ban Tsui, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wheeler M, Oderda GM, Ashburn MA, Lipman AG. Adverse events associated with postoperative opioid analgesia: a systematic review. J Pain. 2002 Jun;3(3):159-80. doi: 10.1054/jpai.2002.123652. No abstract available. PMID 14622770
- [Background] Zhu F, Lee A, Chee YE. Fast-track cardiac care for adult cardiac surgical patients. Cochrane Database Syst Rev. 2012 Oct 17;10:CD003587. doi: 10.1002/14651858.CD003587.pub2. PMID 23076899
- [Background] Baikoussis NG, Papakonstantinou NA, Verra C, Kakouris G, Chounti M, Hountis P, Dedeilias P, Argiriou M. Mechanisms of oxidative stress and myocardial protection during open-heart surgery. Ann Card Anaesth. 2015 Oct-Dec;18(4):555-64. doi: 10.4103/0971-9784.166465. PMID 26440242
- [Background] Giomarelli P, Scolletta S, Borrelli E, Biagioli B. Myocardial and lung injury after cardiopulmonary bypass: role of interleukin (IL)-10. Ann Thorac Surg. 2003 Jul;76(1):117-23. doi: 10.1016/s0003-4975(03)00194-2. PMID 12842524
- [Background] Fragiadakis GK, Gaudilliere B, Ganio EA, Aghaeepour N, Tingle M, Nolan GP, Angst MS. Patient-specific Immune States before Surgery Are Strong Correlates of Surgical Recovery. Anesthesiology. 2015 Dec;123(6):1241-55. doi: 10.1097/ALN.0000000000000887. PMID 26655308
- [Background] Gaudilliere B, Fragiadakis GK, Bruggner RV, Nicolau M, Finck R, Tingle M, Silva J, Ganio EA, Yeh CG, Maloney WJ, Huddleston JI, Goodman SB, Davis MM, Bendall SC, Fantl WJ, Angst MS, Nolan GP. Clinical recovery from surgery correlates with single-cell immune signatures. Sci Transl Med. 2014 Sep 24;6(255):255ra131. doi: 10.1126/scitranslmed.3009701. PMID 25253674
- [Background] Eljezi V, D'Ostrevy N. Local Anesthetic Diffusion of Bilateral Sternal Block After Cardiac Surgery. Reg Anesth Pain Med. 2017 May/Jun;42(3):418-419. doi: 10.1097/AAP.0000000000000577. No abstract available. PMID 28419054
- [Background] Chaudhary V, Chauhan S, Choudhury M, Kiran U, Vasdev S, Talwar S. Parasternal intercostal block with ropivacaine for postoperative analgesia in pediatric patients undergoing cardiac surgery: a double-blind, randomized, controlled study. J Cardiothorac Vasc Anesth. 2012 Jun;26(3):439-42. doi: 10.1053/j.jvca.2011.10.012. Epub 2011 Dec 16. PMID 22176767
- [Background] Olivier JF, Bracco D, Nguyen P, Le N, Noiseux N, Hemmerling T; Perioperative Cardiac Surgery Research Group (PeriCARG). A novel approach for pain management in cardiac surgery via median sternotomy: bilateral single-shot paravertebral blocks. Heart Surg Forum. 2007;10(5):E357-62. doi: 10.1532/HSF98.20071082. PMID 17855198
- [Background] Canto M, Sanchez MJ, Casas MA, Bataller ML. Bilateral paravertebral blockade for conventional cardiac surgery. Anaesthesia. 2003 Apr;58(4):365-70. doi: 10.1046/j.1365-2044.2003.03082_2.x. PMID 12688271
- [Background] Lockwood GG, Cabreros L, Banach D, Punjabi PP. Continuous bilateral thoracic paravertebral blockade for analgesia after cardiac surgery: a randomised, controlled trial. Perfusion. 2017 Oct;32(7):591-597. doi: 10.1177/0267659117715507. Epub 2017 Jun 7. PMID 28592166
- [Background] Svircevic V, Nierich AP, Moons KG, Diephuis JC, Ennema JJ, Brandon Bravo Bruinsma GJ, Kalkman CJ, van Dijk D. Thoracic epidural anesthesia for cardiac surgery: a randomized trial. Anesthesiology. 2011 Feb;114(2):262-70. doi: 10.1097/ALN.0b013e318201d2de. PMID 21239976
- [Background] Chakravarthy M, Thimmangowda P, Krishnamurthy J, Nadiminti S, Jawali V. Thoracic epidural anesthesia in cardiac surgical patients: a prospective audit of 2,113 cases. J Cardiothorac Vasc Anesth. 2005 Feb;19(1):44-8. doi: 10.1053/j.jvca.2004.11.008. PMID 15747268
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] Kose HC, Kose SG, Thomas DT. Lumbar versus thoracic erector spinae plane block: Similar nomenclature, different mechanism of action. J Clin Anesth. 2018 Aug;48:1. doi: 10.1016/j.jclinane.2018.03.026. Epub 2018 Apr 9. No abstract available. PMID 29649625
- [Background] Wong J, Navaratnam M, Boltz G, Maeda K, Ramamurthi RJ, Tsui BCH. Bilateral continuous erector spinae plane blocks for sternotomy in a pediatric cardiac patient. J Clin Anesth. 2018 Jun;47:82-83. doi: 10.1016/j.jclinane.2018.03.020. Epub 2018 Apr 6. No abstract available. PMID 29631111
- [Background] Tsui BCH, Navaratnam M, Boltz G, Maeda K, Caruso TJ. Bilateral automatized intermittent bolus erector spinae plane analgesic blocks for sternotomy in a cardiac patient who underwent cardiopulmonary bypass: A new era of Cardiac Regional Anesthesia. J Clin Anesth. 2018 Aug;48:9-10. doi: 10.1016/j.jclinane.2018.04.005. Epub 2018 May 26. No abstract available. PMID 29684728
- [Background] Kain ZN, Fitch JC, Kirsch JR, Mets B, Pearl RG. Future of anesthesiology is perioperative medicine: a call for action. Anesthesiology. 2015 Jun;122(6):1192-5. doi: 10.1097/ALN.0000000000000680. No abstract available. PMID 25886775